CLINICAL TRIAL: NCT04305080
Title: The Effect of Anodic Oxidation of Implant Abutment Collar on the Peri-implant Soft Tissue Health (Randomized Controlled Clinical Trial)
Brief Title: Effect of Anodic Oxidation of Implant Abutment Collar on the Peri-implant Soft Tissue Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nourhan M.Aly (Other)
Collaborators: Alexandria University (Other)
Responsible Party: Sponsor-Investigator, Nourhan M.Aly, Instructor of Dental Public Health and Statistician, University of Alexandria
Organization: University of Alexandria (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Anodic oxidation
Record Dates: First submitted 2020-03-09; First posted 2020-03-12 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Dental Implants

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anodic Oxidation of implant abutment (Experimental)
  Interventions: Other: Anodic oxidation
- Untreated implant abutment (Sham Comparator)
  Interventions: Other: Untreated abutment

INTERVENTIONS:
Other: Anodic oxidation — Abutments will undergo anodic oxidation process after etching with Hydrofluoric acid & Nitric acid mixture for 10 minutes for debridement in a bath of distilled water with citric acid for 5 minutes to turn the abutment collar into pink color. The stainless steel plate will be connected to the cathode (-) and titanium abutments will be connected to the anode (+) end of the DC Power Supply. After then abutments will be left in distilled water for 10 minutes and sterilized before insertion in patient mouth.
  Arms: Anodic Oxidation of implant abutment
Other: Untreated abutment — Abutment will be left untreated with its gray color.
  Arms: Untreated implant abutment

SUMMARY:
This research aims to evaluate the effect of anodic oxidation of implant abutment collar on the peri-implant soft tissue health.

DETAILED DESCRIPTION:
A randomized controlled clinical trial will be implemented on 10 implant abutments in five patients, each having 2 dental implants in the same quadrant. Abutments with standard silver collars will be divided into two groups: Group 1 (test group) will undergo anodic oxidation of the abutment collar changing it into pink color. Group 2 (control group) untreated abutments.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients with good oral hygiene.
* Having two inserted dental implants in the same quadrant with healing abutments.
* Implants with at least 1 mm peri-implant soft tissue height.

Exclusion Criteria:

* Patients with systemic conditions interfering with soft tissue health.
* Heavy smoking.
* Patients with inflamed gingival tissue or bad oral hygiene.
* Diseased gingival tissue that needs periodontal treatment.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2019-10-20 (Actual); Primary Completion 2020-08-15 (Actual); Study Completion 2020-10-07 (Actual)

PRIMARY OUTCOMES:
Pink aesthetic score | baseline
  Each variable will be assessed using the 0-2 scoring; with 2 being the highest score and 0 the lowest score. The highest possible score is 14 reflecting a peri-implant tissue that is most similar to the soft tissues of the reference tooth. The mesial and distal papillae will be assessed as complete, incomplete, or absent.
Pink aesthetic score | 6 months
  Each variable will be assessed using the 0-2 scoring; with 2 being the highest score and 0 the lowest score. The highest possible score is 14 reflecting a peri-implant tissue that is most similar to the soft tissues of the reference tooth. The mesial and distal papillae will be assessed as complete, incomplete, or absent.
Plaque index (Silness-Löe Index) | baseline
  This will be assessed on 4 surfaces of 6 index teeth. Each of the four surfaces of the teeth (buccal, lingual, mesial and distal) is given a score from 0-3. The scores from the four areas of the tooth are added and divided by four in order to give the plaque index for the tooth with the following scores and criteria. 0:No plaque, 1: A film of plaque adhering to the free gingival margin and adjacent area of the tooth. The plaque may be seen in situ only after application of disclosing solution or by using the probe on the tooth surface.
  2: Moderate accumulation of soft deposit s within the gingival pocket, or the tooth and gingival margin which can be seen with the naked eye. 3: Abundance of soft matter within the gingival pocket and/or on the tooth and gingival margin.
Plaque index (Silness-Löe Index) | 6 months
  This will be assessed on 4 surfaces of 6 index teeth. Each of the four surfaces of the teeth (buccal, lingual, mesial and distal) is given a score from 0-3. The scores from the four areas of the tooth are added and divided by four in order to give the plaque index for the tooth with the following scores and criteria. 0:No plaque, 1: A film of plaque adhering to the free gingival margin and adjacent area of the tooth. The plaque may be seen in situ only after application of disclosing solution or by using the probe on the tooth surface.
  2: Moderate accumulation of soft deposit s within the gingival pocket, or the tooth and gingival margin which can be seen with the naked eye. 3: Abundance of soft matter within the gingival pocket and/or on the tooth and gingival margin.
Probing depth | baseline
  measured using Michigan "O" probe with William's calibrations ((Hu-Friedy, Chicago, IL, USA) at 6 points around the tooth
Probing depth | 6 months
  measured using Michigan "O" probe with William's calibrations ((Hu-Friedy, Chicago, IL, USA) at 6 points around the tooth
Bleeding on probing | baseline
  measured using Michigan "O" probe with William's calibrations ((Hu-Friedy, Chicago, IL, USA) at 6 points around the tooth
Bleeding on probing | 6 months
  measured using Michigan "O" probe with William's calibrations ((Hu-Friedy, Chicago, IL, USA) at 6 points around the tooth

CONTACTS AND LOCATIONS:
Overall Officials: Khaled Farrag, BDS, Principal Investigator — Faculty of Dentistry, Alexandria University, Egypt; Moataz Khamis, PhD, Study Chair — Faculty of Dentistry, Alexandria University, Egypt
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt

REFERENCES:
- [Background] Gehrke P, Lobert M, Dhom G. Reproducibility of the pink esthetic score--rating soft tissue esthetics around single-implant restorations with regard to dental observer specialization. J Esthet Restor Dent. 2008;20(6):375-84; discussion 385. doi: 10.1111/j.1708-8240.2008.00212.x. PMID 19120783
- [Background] Diamanti MV, Del Curto B, Pedeferri M. Anodic oxidation of titanium: from technical aspects to biomedical applications. J Appl Biomater Biomech. 2011 Jan-Apr;9(1):55-69. doi: 10.5301/JABB.2011.7429. PMID 21607937
- [Background] Furhauser R, Florescu D, Benesch T, Haas R, Mailath G, Watzek G. Evaluation of soft tissue around single-tooth implant crowns: the pink esthetic score. Clin Oral Implants Res. 2005 Dec;16(6):639-44. doi: 10.1111/j.1600-0501.2005.01193.x. PMID 16307569